CLINICAL TRIAL: NCT02025036
Title: Three-arm Phase III Trial Comparing Radiotherapy With Different Chemotherapy Regimens for Esophageal Cancer
Brief Title: Chemoradiotherapy of Capecitabine With or Without Oxaliplatin Versus Cisplatin-5-FU for Esophageal Squamous Cancer
Acronym: CRTCOESC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Collaborators: Luoyang Central Hospital (Other); Military 150 Hospital (Unknown); Anyang Cancer Hospital (Unknown); Nanyang Central Hospital (Other); Henan Oncology Hospital (Unknown); The First Affiliated Hospital of Xinyang Medical College (Unknown); Sanmenxia Central Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstHenanUST
Record Dates: First submitted 2013-11-17; First posted 2013-12-31 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Stage III Esophageal Squamous Cell Carcinoma; Stage II Esophageal Squamous Cell Carcinoma
Keywords: Chemoradiotherapy， Esophageal Squamous Cancer
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Capecitabine-oxaliplatin-radiotherapy (Experimental): oxaliplatin：65mg/m2，d1，8，22, 29,I.V.or d1, 8, 22, 29, 43, 50, 64, 71,I.V.plus,capecitabine: 625mg/m2, bid d1-5; q1w, po,6 weeks or 12 weeks in total.
  radiotherapy： 50-50.4Gy ，1.8-2 Gy/d，5d/w.
  Interventions: Drug: Capecitabine(Aibin); Drug: Oxaliplatin(Aiheng); Radiation: Radiotherapy
- cisplatin with 5-FU and radiotherapy (Active Comparator): cisplatin: 75mg/m2 d1，29 or d1, 29, 57, 85, 5-Fu：750mg/m2 CIV24h d1-4，d29-32 or d1-4，d29-32, d57-60, d85-88.
  radiotherapy： 50-50.4Gy ，1.8-2 Gy/d，5d/w.
  Interventions: Radiation: Radiotherapy
- Capecitabine and radiotherapy (Experimental): capecitabine: 625mg/m2, bid d1-5; q1w, po,6 weeks or 12 weeks in total, radiotherapy： 50-50.4Gy ，1.8-2 Gy/d，5d/w.
  Interventions: Drug: Capecitabine(Aibin); Radiation: Radiotherapy

INTERVENTIONS:
Drug: Capecitabine(Aibin) — capecitabine(Aibin)：625mg/m2, bid d1-5; q1w, po,5 weeks in total
  Other Names: Aibin
  Arms: Capecitabine and radiotherapy; Capecitabine-oxaliplatin-radiotherapy
Drug: Oxaliplatin(Aiheng) — Oxaliplatin(Aiheng)：65mg/m2，d1，8, 22, 29,I.V.
  Other Names: Aiheng
  Arms: Capecitabine-oxaliplatin-radiotherapy
Radiation: Radiotherapy — concurrent radiotherapy： 50Gy in total，2 Gy/d，5d/w，Until disease progression or unacceptable toxicity
  Other Names: Radiation Therapy

SUMMARY:
A three-arm Phase III trial was started in Oct. 2014. Definitive chemoradiotherapy with cisplatin plus 5-fluorouracil is the standard in Western countries in esophagus cancer. But in China because of its toxic reaction, most of patients stop the halfway. Because low toxicity, the chemotherapy regimen of capecitabine with or without oxaliplatin are widely used in clinical.

The purpose of this study is to confirm the difference of Capecitabine plus with or without oxaliplatin over cisplatin plus 5-fluorouracil with definitive chemoradiotherapy for esophagus squamous cell carcinoma. A total of 249 patients will be accrued from China within 2 years. The primary endpoints are grade 3-5 AEs and overall survival and the secondary endpoints include progression-free survival, response rate, pathologic complete response rate.

DETAILED DESCRIPTION:
We plan to recruit the patients who were pathologically confirmed with esophageal squamous cell carcinoma from the Oct 2014. The patients will be divided into three groups.Experimental group 1 : single drug Capecitabine and concurrent radiotherapy.Experimental group 2: Capecitabine plus oxaliplatin and concurrent radiotherapy. Control group:cisplatin plus 5-fluorouracil and concurrent radiotherapy. To evaluate the adverse events and the overall survival of the three group. Also observe the patient's progression-free survival, response rate, pathologic complete response rate.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75years old
* Histologically proven squamous cell carcinoma of the esophagus the tumor was in T2-4N0-2M0
* The patients have not received the surgery or chemo-radiotherapy.
* Hb≥80g/L, absolute neutrophil count ≥1.5×109/L, Plt≥90×109/L,
* ALT、AST≤2.5*N,Cr≤1.5*N.
* performance status score 0-2

Exclusion Criteria:

* pregnant, lactating women
* Oxaliplatin or fluorouracil Allergy or metabolic disorders
* Radiotherapy contraindications
* History of organ transplantation
* Brain metastasis
* The peripheral nervous system disorders
* Severe infection
* Oral capecitabine who have difficulty with,such as dysphagia,The activities of digestive ulcer, Gastrointestinal bleeding
* Severe chronic diseases, such as, hepatopathy, nephropathy, respiratory disease,high blood pressure, diabetes.
* Other malignant tumor in recent 5 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Grade 3/5 acute toxicities | 90 days
  Grade 3/5 acute toxicities occurred during or within 90 days after RT
OS-2 year | 2 years
  Overall Survival rate in 2 year from Randomization

SECONDARY OUTCOMES:
PFS-2 year | 2 years
  Progression Free Survival rate in 2 year from Randomization
overall remission rate, ORR | 16 weeks
  overall remission rate after CRT
quality of life, Qol | 16 weeks
  quality of life evaluation
pathologic complete response rate | 16 weeks
  pathologic complete response rate confirmed by gastroscope biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, M.D Ph.D, Study Chair — The First Affiliated Hospital of Henan University of Science and Technology; Tanyou Shan, M.D M.S, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Xiaoshan Feng, M.D Ph.D, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Jiachun Sun, M.D Ph.D, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Xinshuai Wang, M.D Ph.D, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Guoqiang Kong, M.D M.S, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Xiaozhi Yuan, M.D M.S, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Ruinuo Jia, M.D Ph.D, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Dan Zhou, M.D M.S, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Jing Ren, M.D M.S, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Ruina Yang, M.D M.S, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Dan Wang, M.D M.S, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Wei Wang, M.D M.S, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Yali Zhang, M.D M.S, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Yongxuan Liu, M.D M.S, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Weijiao Yin, M.D M.S, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Shiyuan Song, M.D M.S, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Guobao Zheng, M.D Ph.D, Principal Investigator — No. 150 Central Hospital of the Chinese People Liberation Army; Daoke Yang, M.D M.S, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Jianhua Wang, M.D Ph.D, Principal Investigator — Henan Tumor Hospital; Fuyou Zhou, M.D Ph.D, Principal Investigator — Anyang Tumour Hospital of Henan province; Nengchao Wang, M.D M.S, Principal Investigator — Anyang Tumour Hospital of Henan province; Anping Zheng, M.D M.S, Principal Investigator — Anyang Tumour Hospital of Henan province; Zhanhui Miao, M.D M.S, Principal Investigator — Affiliated Hospital of Xinxiang Medical University, Henan province; Ruiwen Zhang, M.D M.S, Principal Investigator — Xinxiang Central Hospital of Henan province
Locations (1):
- The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park JW, Kim JH, Choi EK, Lee SW, Yoon SM, Song SY, Lee YS, Kim SB, Park SI, Ahn SD. Prognosis of esophageal cancer patients with pathologic complete response after preoperative concurrent chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):691-7. doi: 10.1016/j.ijrobp.2010.06.041. Epub 2010 Oct 1. PMID 20888705
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Blum MA, Taketa T, Sudo K, Wadhwa R, Skinner HD, Ajani JA. Chemoradiation for esophageal cancer. Thorac Surg Clin. 2013 Nov;23(4):551-8. doi: 10.1016/j.thorsurg.2013.07.006. PMID 24199704
- [Background] Conroy T, Galais MP, Raoul JL, Bouche O, Gourgou-Bourgade S, Douillard JY, Etienne PL, Boige V, Martel-Lafay I, Michel P, Llacer-Moscardo C, Francois E, Crehange G, Abdelghani MB, Juzyna B, Bedenne L, Adenis A; Federation Francophone de Cancerologie Digestive and UNICANCER-GI Group. Definitive chemoradiotherapy with FOLFOX versus fluorouracil and cisplatin in patients with oesophageal cancer (PRODIGE5/ACCORD17): final results of a randomised, phase 2/3 trial. Lancet Oncol. 2014 Mar;15(3):305-14. doi: 10.1016/S1470-2045(14)70028-2. Epub 2014 Feb 18. PMID 24556041
- [Background] Kato K, Muro K, Minashi K, Ohtsu A, Ishikura S, Boku N, Takiuchi H, Komatsu Y, Miyata Y, Fukuda H; Gastrointestinal Oncology Study Group of the Japan Clinical Oncology Group (JCOG). Phase II study of chemoradiotherapy with 5-fluorouracil and cisplatin for Stage II-III esophageal squamous cell carcinoma: JCOG trial (JCOG 9906). Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):684-90. doi: 10.1016/j.ijrobp.2010.06.033. Epub 2010 Oct 6. PMID 20932658
- [Background] Kato K, Nakajima TE, Ito Y, Katada C, Ishiyama H, Tokunaga SY, Tanaka M, Hironaka S, Hashimoto T, Ura T, Kodaira T, Yoshimura K. Phase II study of concurrent chemoradiotherapy at the dose of 50.4 Gy with elective nodal irradiation for Stage II-III esophageal carcinoma. Jpn J Clin Oncol. 2013 Jun;43(6):608-15. doi: 10.1093/jjco/hyt048. Epub 2013 Apr 12. PMID 23585687
- [Background] Lee SJ, Ahn BM, Kim JG, Sohn SK, Chae YS, Moon JH, Lee EB, Kim JC, Park IK, Jeon SW. Definitive chemoradiotherapy with capecitabine and cisplatin in patients with esophageal cancer: a pilot study. J Korean Med Sci. 2009 Feb;24(1):120-5. doi: 10.3346/jkms.2009.24.1.120. Epub 2009 Feb 28. PMID 19270824
- [Background] Xing L, Liang Y, Zhang J, Wu P, Xu D, Liu F, Yu X, Jiang Z, Song X, Zang Q, Wang W. Definitive chemoradiotherapy with capecitabine and cisplatin for elder patients with locally advanced squamous cell esophageal cancer. J Cancer Res Clin Oncol. 2014 May;140(5):867-72. doi: 10.1007/s00432-014-1615-5. Epub 2014 Mar 1. PMID 24578238
- [Derived] Jia R, Shan T, Zheng A, Zhang Y, Lu P, Zhang G, Wang F, Xu Z, Zheng G, Tang D, Zhang W, Li W, Li R, Guo Y, Liu L, Luo X, Zheng Y, Chang Z, Wang Q, Wang X, Yuan X, Kong G, Li S, Yang R, Zhou D, Ren J, Yin W, Li J, Zhang J, Wang Z, Sheng M, Xu B, Li L, Liu X, Lu Z, Wan L, Zhou F, Gao S. Capecitabine or Capecitabine Plus Oxaliplatin Versus Fluorouracil Plus Cisplatin in Definitive Concurrent Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma (CRTCOESC): A Multicenter, Randomized, Open-Label, Phase 3 Trial. J Clin Oncol. 2024 Jul 10;42(20):2436-2445. doi: 10.1200/JCO.23.02009. Epub 2024 May 6. PMID 38710003